CLINICAL TRIAL: NCT04875806
Title: A Phase 1/2, Open-Label, Dose-Escalation, Safety and Tolerability Study of NC762 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Safety and Tolerability Study of NC762 in Subjects With Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the limited activity in Phase 1, NextCure decided to discontinue development of the anti-B7-H4 antibody monotherapy trial (NC762-01) to move forward with a prioritized B7-H4 ADC program.
Sponsor: NextCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NC762-01
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Advanced or Metastatic Solid Tumors; Ovarian Cancer; Non-small Cell Lung Cancer; Breast Cancer
Keywords: Advanced Cancer; Metastatic Cancer; NC762; Solid Tumor; Immunotherapy; PK; Ovarian Cancer; Lung Cancer; Breast Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Neoplasm Metastasis; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1 will utilize a 3 + 3 design to explore escalating dose levels. Phase 2 Dose Expansion will further evaluate the safety, tolerability, preliminary efficacy, and PK/PD activity of NC762 at the RP2D utilizing a Simon 2-stage design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 0.5mg/kg NC762 (Experimental): Subjects received NC762 IV at 0.5mg/kg Q2W until disease progression, withdraw of consent, or intolerable toxicity (whichever comes first).
  Interventions: Drug: NC762
- 1.5mg/kg NC762 (Experimental): Subjects received NC762 IV at 1.5mg/kg Q2W until disease progression, withdraw of consent, or intolerable toxicity (whichever comes first).
  Interventions: Drug: NC762
- 5mg/kg NC762 (Experimental): Subjects received NC762 IV at 5mg/kg Q2W until disease progression, withdraw of consent, or intolerable toxicity (whichever comes first).
  Interventions: Drug: NC762
- 10mg/kg NC762 (Experimental): Subjects received NC762 IV at 10mg/kg Q2W until disease progression, withdraw of consent, or intolerable toxicity (whichever comes first).
  Interventions: Drug: NC762
- 20mg/kg NC762 (Experimental): Subjects received NC762 IV at 20mg/kg Q2W until disease progression, withdraw of consent, or intolerable toxicity (whichever comes first).
  Interventions: Drug: NC762

INTERVENTIONS:
Drug: NC762 — NC762 is an experimental antibody drug that may make the immune response more active against cancer

SUMMARY:
This research study is studying a new drug, NC762, as a possible treatment for advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or older.
* Willingness to provide written informed consent for the study.
* ECOG performance status 0 to 1.
* Locally advanced or metastatic disease; locally advanced disease must not be amenable to resection with curative intent.
* Subjects who have disease progression after treatment with available therapies that are known to confer clinical benefit, or who are intolerant to treatment, or who refuse standard treatment. Note: There is no limit to the number of prior treatment regimens.
* Presence of measurable disease based on RECIST v1.1. Tumor lesions situated in a previously irradiated area, or in an area subjected to other locoregional therapy, are not considered measurable unless there has been demonstrated progression in the lesion.
* Phase 1a Dose Escalation (optional), Phase 1b Safety Expansion, and Phase 2 (mandatory): Willingness to undergo pretreatment and on-treatment tumor biopsies (core or excisional).
* Female subjects of childbearing potential (defined as women who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy and are not postmenopausal, defined as ≥ 12 months of amenorrhea) and non-sterilized male subjects of childbearing potential must agree to take appropriate precautions to avoid pregnancy or fathering children (with at least 99% certainty) from screening through 90 days after the last dose of study drug. Females of child-bearing potential must have a negative serum pregnancy test at screening.

Exclusion Criteria:

* Inability to comprehend or unwilling to sign the ICF.
* Laboratory and medical history parameters not within the protocol-defined range.

  1. Absolute neutrophil count < 1.5 × 10^9/L.
  2. Platelets < 100 × 10^9/L.
  3. Hemoglobin < 9 g/dL or < 5.6 mmol/L.
  4. Serum creatinine > 1.5 × institutional upper limit of normal (ULN) and measured or calculated creatinine clearance < 50 mL/min for subjects with creatinine levels > 1.5 × institutional ULN.
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥ 2.5 × ULN. With the following exceptions: subjects with documented liver metastases AST and/or ALT ≤ 5 × ULN. Patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 ×ULN.
  6. Total bilirubin ≥ 1.5 × ULN.
  7. International normalized ratio (INR) or prothrombin time (PT) > 1.5 × ULN; Activated partial thromboplastin time (aPTT) > 1.5 × ULN, except for subjects on anticoagulation.
* Transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 7 days before the first administration of study drug.
* Receipt of anticancer medications or investigational drugs within the following intervals before the first administration of study drug:

  1. ≤ 14 days for chemotherapy, targeted small molecule therapy, hormonal therapy or radiation therapy. Subjects must not have had radiation pneumonitis because of a treatment. A 1-week washout is permitted for palliative radiation to non-central nervous system (CNS) disease with medical monitor approval.
  2. ≤ 28 days for prior immunotherapy or persistence of active cellular therapy (e.g., chimeric antigen receptor T cell therapy; other cellular therapies must be discussed with the medical monitor to determine eligibility).
  3. ≤ 28 days for a prior mAb used for anticancer therapy except for denosumab.
  4. ≤ 7 days for immune-suppressive-based treatment for any reason.
  5. ≤ 28 days or 5 half-lives, t½, (whichever is longer) before the first dose for all other investigational study drugs or devices. For investigational agents with long half-lives (e.g., > 5 days), enrollment before the fifth t½ requires medical monitor approval.
  6. ≤ 14 days for a COVID-19 vaccine. Note: For 2-dose vaccines, subjects must wait at least 14 days after administration of the 2nd dose of the vaccine prior to receiving the first dose of the study drug.
* Has not recovered to ≤ Grade 1 from toxic effects of prior therapy (including prior immunotherapy and radiation therapy) and/or complications from prior surgical intervention before starting therapy.
* Receipt of a live vaccine within 30 days of planned start of study therapy.
* Active autoimmune disease that required systemic treatment in the past (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).
* Known active CNS metastases and/or carcinomatous meningitis.
* Known concurrent malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry.
* Evidence of active, noninfectious pneumonitis or history of interstitial lung disease.
* Documented known activating or driver mutations (i.e. EGFR mutations/amplification, BRAF mutations, ALK alterations, etc.) which have not been previously treated with a standard of care targeted therapy.
* Subjects with screening QTc interval > 470 milliseconds (corrected by Fridericia) are excluded.
* Uncontrolled systemic fungal, bacterial, viral, or other infection despite appropriate anti-infection treatment.
* Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV), unless the hepatitis is considered to be cured.
* Known history of HIV (HIV 1 or HIV 2 antibodies).
* Known allergy or reaction to any component of study drug or formulation components.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 90 days after the last dose of study treatment.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han Myint, MD, Study Director — NextCure, Inc.
Locations (8):
- United States (8):
  - Yale Cancer Center, New Haven, Connecticut
  - The University of Chicago Medicine and Biological Sciences, Chicago, Illinois
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.5mg/kg NC762 | 1.5mg/kg NC762 | 5mg/kg NC762 | 10mg/kg NC762 | 20mg/kg NC762
Started | 4 | 4 | 3 | 11 | 18
Completed | 3 | 2 | 2 | 5 | 13
Not Completed | 1 | 2 | 1 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5mg/kg NC762 | 1.5mg/kg NC762 | 5mg/kg NC762 | 10mg/kg NC762 | 20mg/kg NC762 | Total
Number analyzed (Participants) | 4 | 4 | 3 | 11 | 18 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (4.03) | 74.0 (8.76) | 74.3 (3.21) | 61.5 (13.13) | 57.0 (13.55) | 60.4 (13.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 7 | 18 | 28
  Male | 3 | 3 | 2 | 4 | 0 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 4 | 3 | 11 | 17 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 3 | 4
  White | 3 | 4 | 2 | 11 | 14 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 3 | 11 | 18 | 40
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Population: One participant in 10mg/kg cohort did not have baseline height collected, therefore baseline BMI could not be calculated.
  kg/m2
    number analyzed (Participants) | 4 | 4 | 3 | 10 | 18 | 39
    (all) | 22.693 (4.6895) | 29.365 (4.2638) | 26.543 (4.5224) | 26.366 (5.5265) | 25.937 (6.0424) | 26.113 (5.4960)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events as Assessed by CTCAE v5.0
Description: Frequency, duration, and severity of treatment-emergent adverse events (AEs)
Time Frame: From enrollment through up to 90 days after end of treatment, an average of 1 year
Population: The Safety Analysis Set (SAS) will include all the subjects who receive any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5mg/kg NC762 | 1.5mg/kg NC762 | 5mg/kg NC762 | 10mg/kg NC762 | 20mg/kg NC762
Number analyzed (Participants) | 4 | 4 | 3 | 11 | 18
Participants | 4 | 3 | 3 | 11 | 18

2. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: To assess antitumor activity/efficacy by evaluating objective response rate (ORR), defined as the percentage of participants who experienced a complete response (CR; disappearance of all target lesions) or a partial response (PR; at least a 30% decrease in the sum of diameters of target lesions) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Time Frame: Approximately 1 year
Population: The full analysis set (FAS) includes all subjects enrolled in the study who received at least one full dose of NC762
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5mg/kg NC762 | 1.5mg/kg NC762 | 5mg/kg NC762 | 10mg/kg NC762 | 20mg/kg NC762
Number analyzed (Participants) | 4 | 4 | 3 | 11 | 18
Participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Duration of Response (DoR) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: To assess antitumor activity/efficacy by evaluating duration of response (DoR), defined as the time from the first documented complete response or partial response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 to the first documented progressive disease or death due to any cause, whichever occurs first. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Approximately 1 year
Population: The full analysis set (FAS) includes all subjects enrolled in the study who received at least one full dose of NC762
Measure: Median (99% Confidence Interval); unit: months
Arm/Group | 0.5mg/kg NC762 | 1.5mg/kg NC762 | 5mg/kg NC762 | 10mg/kg NC762 | 20mg/kg NC762
Number analyzed (Participants) | 4 | 4 | 3 | 11 | 18
months | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events.

4. Secondary Outcome: Disease Control Rate (DCR) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: To assess antitumor activity/efficacy by evaluating disease control rate (DCR), defined as the proportion of participants in whom a documented complete response, partial response, or stable disease is observed as the best overall response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Time Frame: Approximately 1 year
Population: The FAS includes all subjects enrolled in the study who received at least one full dose of NC762
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5mg/kg NC762 | 1.5mg/kg NC762 | 5mg/kg NC762 | 10mg/kg NC762 | 20mg/kg NC762
Number analyzed (Participants) | 4 | 4 | 3 | 11 | 18
Participants | 2 | 3 | 2 | 3 | 6

5. Secondary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: To evaluate progression-free survival (PFS), defined as the time from the first dose of NC762 to the first occurrence of documented progressive disease or death due to any cause, whichever occurs first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Approximately 1 year
Population: The FAS includes all subjects enrolled in the study who received at least one full dose of NC762
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | 0.5mg/kg NC762 | 1.5mg/kg NC762 | 5mg/kg NC762 | 10mg/kg NC762 | 20mg/kg NC762
Number analyzed (Participants) | 4 | 4 | 3 | 11 | 18
weeks | 12.07 [7.14 to NA] — The upper limit of the confidence interval were not estimable due to limited number of participants with events. | 13.00 [7.86 to NA] — The upper limit of the confidence interval were not estimable due to limited number of participants with events. | 33.29 [6.29 to NA] — The upper limit of the confidence interval were not estimable due to limited number of participants with events. | 7.43 [6.29 to NA] — The upper limit of the confidence interval were not estimable due to limited number of participants with events. | 7.57 [5.43 to 15.43]

6. Secondary Outcome: Overall Survival (OS)
Description: To evaluate overall survival (OS), defined as the time from the first dose of NC762 to death due to any cause.
Time Frame: Approximately 1 year
Population: The full analysis set (FAS) includes all subjects enrolled in the study who received at least one full dose of NC762
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 0.5mg/kg NC762 | 1.5mg/kg NC762 | 5mg/kg NC762 | 10mg/kg NC762 | 20mg/kg NC762
Number analyzed (Participants) | 4 | 4 | 3 | 11 | 18
months | NA [2.86 to NA] — The median and upper limit of the confidence interval were not estimable due to limited number of participants with event. | 15.74 [NA to NA] — Confidence intervals were not estimable as survival curve hasn't reached a point where meaningful lower/upper limits can be estimated, due to limited follow-up and/or censoring. | 7.66 [2.23 to NA] — The upper limit of the confidence interval was not estimable due to limited number of participants with event. | NA [2.92 to NA] — The median and upper limit of the confidence interval were not estimable due to limited number of participants with event. | 7.92 [1.64 to NA] — The upper limit of the confidence interval was not estimable due to limited number of participants with event.

7. Secondary Outcome: Maximum Serum Concentration (Cmax) of NC762
Description: To evaluate the Maximum Serum Concentration (Cmax) of NC762
Time Frame: Days 1, 2, 3, and 8 of Cycles 1 and 5. Each cycle is 14 days.
Population: The PK analysis set (PAS) will include all the subjects whose blood samples are collected for PK analysis.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | 0.5mg/kg NC762 | 1.5mg/kg NC762 | 5mg/kg NC762 | 10mg/kg NC762 | 20mg/kg NC762
Number analyzed (Participants) | 4 | 4 | 2 | 11 | 16
ug/mL
  Cycle 1 | 11.2 (2.62) | 18.5 (4.98) | 119 (0.707) | 227 (69.6) | 440 (102)
  Cycle 5: number analyzed (Participants) | 2 | 3 | 1 | 3 | 5
  Cycle 5 | 14.6 (6.08) | 35.8 (6.21) | NA (NA) — Sample size too small (n=1) to calculate Mean and Standard Deviation at this visit. For each PK parameter, if at least 67% of the subjects had properly determined parameters (i.e., non-not reported [NR] and non-flagged), descriptive statistics were calculated. Otherwise, the descriptive statistics were replaced by NA. | 289 (197) | 477 (163)

8. Secondary Outcome: Area Under the Curve (AUC) of NC762
Description: To evaluate the Area Under the Curve (AUC) of NC762
Time Frame: Days 1, 2, 3, and 8 of Cycles 1 and 5. Each cycle is 14 days.
Population: The PK analysis set (PAS) will include all the subjects whose blood samples are collected for PK analysis. AUC from time 0 to the last measurable concentration.
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | 0.5mg/kg NC762 | 1.5mg/kg NC762 | 5mg/kg NC762 | 10mg/kg NC762 | 20mg/kg NC762
Number analyzed (Participants) | 4 | 4 | 2 | 11 | 16
h*ug/mL
  Cycle 1 | 1170 (439) | 2130 (481) | 13600 (2620) | 28300 (8990) | 47300 (13200)
  Cycle 5: number analyzed (Participants) | 2 | 3 | 1 | 3 | 5
  Cycle 5 | 2040 (976) | 5090 (684) | NA (NA) — Sample size too small (n=1) to calculate Mean and Standard Deviation at this visit. For each PK parameter, if at least 67% of the subjects had properly determined parameters (i.e., non-not reported [NR] and non-flagged), descriptive statistics were calculated. Otherwise, the descriptive statistics were replaced by NA. | 39100 (38000) | 74900 (39100)

9. Secondary Outcome: Half-life (T1/2) of NC762
Description: To evaluate the Half-life (T1/2) of NC762
Time Frame: Days 1, 2, 3, and 8 of Cycles 1 and 5. Each cycle is 14 days.
Population: The PK analysis set (PAS) will include all the subjects whose blood samples are collected for PK analysis. Half-Life Lambda z (h).
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 0.5mg/kg NC762 | 1.5mg/kg NC762 | 5mg/kg NC762 | 10mg/kg NC762 | 20mg/kg NC762
Number analyzed (Participants) | 3 | 2 | 2 | 4 | 8
h
  Cycle 1 | 114 (23.8) | 131 (29) | 129 (12) | 124 (24.5) | 129 (20.5)
  Cycle 5: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1
  Cycle 5 |  |  | NA (NA) — Sample size to small (n=1) to calculate Mean and Standard Deviation at this visit. For each PK parameter, if at least 67% of the subjects had properly determined parameters (i.e., non-not reported [NR] and non-flagged), descriptive statistics were calculated. Otherwise, the descriptive statistics were replaced by NA. | NA (NA) — Sample size to small (n=1) to calculate Mean and Standard Deviation at this visit. For each PK parameter, if at least 67% of the subjects had properly determined parameters (i.e., non-not reported [NR] and non-flagged), descriptive statistics were calculated. Otherwise, the descriptive statistics were replaced by NA. | NA (NA) — Sample size to small (n=1) to calculate Mean and Standard Deviation at this visit. For each PK parameter, if at least 67% of the subjects had properly determined parameters (i.e., non-not reported [NR] and non-flagged), descriptive statistics were calculated. Otherwise, the descriptive statistics were replaced by NA.

ADVERSE EVENTS:
Time Frame: From enrollment through up to 90 days after end of treatment, an average of 1 year.
Description: The severity of AEs will be assessed using NCI CTCAE v5.0 Grades 1 through 4. The NCI CTCAE v5.0 severity of Grade 5 will not be used; AEs resulting in death will be graded accordingly using Grades 1 through 4 and have the outcome noted as fatal.
Arm/Group | 0.5mg/kg NC762 | 1.5mg/kg NC762 | 5mg/kg NC762 | 10mg/kg NC762 | 20mg/kg NC762
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/4 | 2/3 | 2/11 | 9/18
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 1/3 | 1/11 | 11/18
Other Adverse Events (participants affected / at risk) | 4/4 | 3/4 | 3/3 | 11/11 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5mg/kg NC762 (N=4) | 1.5mg/kg NC762 (N=4) | 5mg/kg NC762 (N=3) | 10mg/kg NC762 (N=11) | 20mg/kg NC762 (N=18)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | NA | NA | 1 (1) | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | NA | NA | 0 | 1 (1) | 0
Abdominal Pain (Gastrointestinal disorders) | NA | NA | 0 | 0 | 2 (3)
Encephalopathy (Nervous system disorders) | NA | NA | 0 | 0 | 2 (2)
Sepsis (Infections and infestations) | NA | NA | 0 | 0 | 1 (1)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | NA | NA | 0 | 0 | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | NA | NA | 0 | 0 | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 0 | 1 (1)
Spinal Cord Compression (Nervous system disorders) | NA | NA | 0 | 0 | 1 (1)
Mental Status Change (Psychiatric disorders) | NA | NA | 0 | 0 | 1 (1)
Nausea (Gastrointestinal disorders) | NA | NA | 0 | 0 | 1 (1)
Vomitting (Gastrointestinal disorders) | NA | NA | 0 | 0 | 1 (1)
Pneumonia (Infections and infestations) | NA | NA | 0 | 0 | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | NA | NA | 0 | 0 | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | NA | NA | 0 | 0 | 1 (1)
Ascites (Gastrointestinal disorders) | NA | NA | 0 | 0 | 2 (2)
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 0.5mg/kg NC762 (N=4) | 1.5mg/kg NC762 (N=4) | 5mg/kg NC762 (N=3) | 10mg/kg NC762 (N=11) | 20mg/kg NC762 (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 5 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 3
Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 6
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 4 | 6
Pancreatic mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 6
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 2 | 4 | 5
Feeling jittery (General disorders) | 0 | 0 | 1 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Non-cardia chest pain (General disorders) | 0 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 2
Pain (General disorders) | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Facial bone fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 2 | 1
Ammonia increased (Investigations) | 0 | 0 | 0 | 0 | 1
Amylase increased (Investigations) | 1 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 3 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 1 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 2 | 4
Blood folate decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 2 | 1
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 0 | 2
Carbon dioxide increased (Investigations) | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 2
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 6
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 3
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 2 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 2
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 2 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0/0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0/1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0/0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0/0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0/0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0/0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0/0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0/0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0/0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0/0 | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0/0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0 | 1 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot publish study results before the first multi-center publication. If a multi-center publication is not submitted within 12 months after the end of the study at all sites, or if Sponsor confirms there will be no multi-center publication, the PI may publish study results. However, PI will allow Sponsor at least 30 days to review any publication of study results and Sponsor may request an additional 60 days to review the publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT04875806/Prot_SAP_000.pdf